CLINICAL TRIAL: NCT03775798
Title: Incidence of de Novo Hepatocellular Carcinoma After Direct-acting Antiviral Agents for HCV: a Multicenter Prospective Cohort Study From Latin America.
Brief Title: Incidence of de Novo Hepatocellular Carcinoma After Antiviral Agents for HCV.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, UIC staff, Austral University, Argentina
Other Study IDs: 17-062
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C; Cirrhosis; Antiviral Drug Adverse Reaction
Keywords: direct acting antivirals; hepatitis c; hepatocellular carcinoma
MeSH Terms: conditions — Hepatitis C; Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Direct antiviral agents for hepatitis C — Direct-acting antivirals for hepatitis C

SUMMARY:
The main risk factor for development of hepatocellular carcinoma (HCC) is cirrhosis of any etiology, with an annual incidence risk between 1-6%; currently the leading cause of death in patients with cirrhosis and the 2nd cause of death by cancer worldwide. Chronic hepatitis C (HCV) is the first single cause associated to cirrhosis and HCC in the Western world.

With the advent of new direct antiviral agents (DAA) of chronic HCV infection, virological cure generally exceeds 90% of the cases. Previous studies have shown that the incidence of HCC is lower in patients with virologic cure after treatment with pegINF schemes. However, recently published data, open up more controversy regarding the incidence of HCC after virologic cure with DAA. An increasing incidence of HCC after virologic cure in patients treated with DAA has been observed, opening a paradox yet unexplained.

This project proposes to answer the following clinical research question: in patients with HCV cirrhosis treated with DAA, is there a change in the incidence of hepatocellular carcinoma? To answer this question a prospective longitudinal cohort study of patients with Child Pugh A-B cirrhosis will be held at 3 years minimum follow-up.

A minimum of 210 patients will be included with clinical or histological or non-invasive diagnosis of cirrhosis Child Pugh A or B, with HCV treated with DAA and without hepatocellular carcinoma at the time of enrollment. From this cohort, patients who develop HCC during follow-up will be identified. Routine screening will be done through ultrasound every 6 months in all subjects enrolled and the diagnosis of HCC will be according to recommendations of European and American guidelines.

DETAILED DESCRIPTION:
Name of the study:

INCIDENCE OF HEPATOCELLULAR CARCINOMA IN CIRRHOTIC PATIENTS WITH HEPATITIS C INFECTION, TRETAED WITH DIRECT ANTIVIRAL AGENTS IN LATIN AMERICA: A MULTICENTER PROSPECTIVE COHORT STUDY

With the advent of new direct antiviral agents (DAA) of chronic HCV infection, virological cure generally exceeds 90% of the cases. Previous studies have shown that the incidence of HCC is lower in patients with virologic cure after treatment with pegINF schemes. However, recently published data, open up more controversy regarding the incidence of HCC after virologic cure with DAA. An increasing incidence of HCC after virologic cure in patients treated with DAA has been observed, opening a paradox yet unexplained.

This project proposes to answer the following clinical research question: in patients with HCV cirrhosis treated with DAA, is there a change in the incidence of hepatocellular carcinoma? To answer this question a prospective longitudinal cohort study of patients with Child Pugh A-B cirrhosis will be held at 3 years minimum follow-up.

A minimum of 210 patients will be included with clinical or histological or non-invasive diagnosis of cirrhosis Child Pugh A or B, with HCV treated with DAA and without hepatocellular carcinoma at the time of enrollement. From this cohort, patients who develop HCC during follow-up will be identified. Routine screening will be done through ultrasound every 6 months in all subjects enrolled and the diagnosis of HCC will be according to recommendations of European and American guidelines.

However, preliminary results presented at the last European Congress of Hepatology in Barcelona, Spain, and early published in Journal of Heaptology, open up more controversy regarding the incidence of HCC after virologic cure post DAA. An unexpected higher incidence and recurrence of HCC after treatment with these new drugs has been observed, opening a paradox yet unexplained. Of particular interest then, is to clarify and find if there is a change in the incidence of HCC in HCV cirrhosis after treatment with DAA in our region. It is relevant on the other hand; that this study would be the first longitudinal cohort study evaluating the development of HCC in patients with cirrhosis in Latin America. It is then expected that the results would be extremely important to the medical science from this region.

Clinical Research Question In patients with HCV cirrhosis treated DAA, is there a change in the incidence of hepatocellular carcinoma? Primary Objective To evaluate the incidence of HCC after treatment with DAA in patients with Child Pugh A or B cirrhosis and chronic HCV infection.

Secondary Objectives

Secondary objectives will be related to:

* Incidence of HCC between cured and uncured of HCV with DAA.
* Impact of routine screening on survival in patients with HCC.
* Risk factors for development of hepatocellular carcinoma in patients with HCV treated with DAA.
* Adverse events and incidence of cirrhosis decompensation after DAA.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent (CI) obtained prior to any study specific procedure. Patients should be able to understand written informed and be ready to sign it (ANNEX I).
* Men and women 18 years or older.
* Clinical, histological or non-invasive diagnosis of cirrhosis, according to the American Association for the Study of Liver Diseases, AASLD criteria) [15].
* Child Pugh A or B (ANNEX II). Child Pugh classification should be calculated based on clinical findings and laboratory results during the selection period.
* Chronic Hepatitis C, defined as positive viremia with real time PCR method.
* Current or prior treatment with DAA, including any interferon-free scheme, either in a clinical protocol or treated in the daily practice.
* Co-infection with HIV infection is allowed or Hepatitis B.

Exclusion Criteria:

* • Prior diagnosis of Hepatocellular to treatment with DAA.

  * Previous liver transplantation.
  * Drug addiction, medical, psychological or social problems that may interfere with the patient's participation in the study or evaluation of the results.
  * Pregnancy and/or breastfeeding.
  * Close relationship with the research center; eg close family member of the researcher, dependent (eg employee or student research center that could access study records and data CRF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive non-probability sampling of subjects with clinical, histological or non-invasive diagnosis of cirrhosis, functional status Child Pugh class A or B with chronic HCV infection treated with DAA will be made. On a cohort of patients with these characteristics that meet the following eligibility criteria, a minimum 3-year follow-up will be done.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatocellular carcinoma after direct-acting antivirals for HCV | Three year period
  Cumulative incidence, Hazard ratios (95% CI)

SECONDARY OUTCOMES:
Effectiveness of direct-acting antivirals for HCV | Three year period
  Achievement of RVS
Adverse events after direct-acting antivirals for HCV | Three year period
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Austral, Pilar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Braillon A. Achieving Virological Response in Patients With Hepatitis C Is Only Half Way for Effective Care. Clin Gastroenterol Hepatol. 2021 Mar;19(3):622-623. doi: 10.1016/j.cgh.2020.04.086. Epub 2020 Nov 26. No abstract available. PMID 33248099
- [Derived] Ridruejo E, Pinero F, Mendizabal M, Cheinquer H, Wolff FH, Anders M, Reggiardo V, Ameigeiras B, Palazzo A, Alonso C, Schinoni MI, Zuain MGV, Tanno F, Figueroa S, Santos L, Peralta M, Soza A, Vistarini C, Adrover R, Fernandez N, Perez D, Hernandez N, Estepo C, Bruno A, Descalzi V, Sixto M, Borzi S, Cocozzella D, Zerega A, de Araujo A, Varon A, Silva M; Latin American Liver Research Educational and Awareness Network (LALREAN). Decompensated cirrhosis and liver transplantation negatively impact in DAA treatment response: Real-world experience from HCV-LALREAN cohort. J Med Virol. 2020 Dec;92(12):3545-3555. doi: 10.1002/jmv.26383. Epub 2020 Aug 13. PMID 32749710
- [Derived] Mendizabal M, Pinero F, Ridruejo E, Herz Wolff F, Anders M, Reggiardo V, Ameigeiras B, Palazzo A, Alonso C, Schinoni MI, Videla Zuain MG, Tanno F, Figueroa S, Santos L, Peralta M, Soza A, Vistarini C, Adrover R, Fernandez N, Perez D, Hernandez N, Estepo C, Bruno A, Descalzi V, Sixto M, Borzi S, Cocozzella D, Zerega A, de Araujo A, Varon A, Rubinstein F, Cheinquer H, Silva M; Latin American Liver Research; Educational and Awareness Network (LALREAN). Disease Progression in Patients With Hepatitis C Virus Infection Treated With Direct-Acting Antiviral Agents. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2554-2563.e3. doi: 10.1016/j.cgh.2020.02.044. Epub 2020 Feb 28. PMID 32113892